CLINICAL TRIAL: NCT00147147
Title: Randomized Trial of Adjuvant Chemotherapy With Cisplatin Followed by Oral Fluorouracil (UFT) in Serosa-positive Gastric Cancer (JCOG9206-2)
Brief Title: Randomized Trial of Adjuvant Chemotherapy With Cisplatin Followed by UFT in Serosa-positive Gastric Cancer (JCOG9206-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9206-2; C000000067
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Neoplasm
Keywords: gastric neoplasm; gastrectomy; adjuvant chemotherapy; randomized trial; T3 and T4 carcinoma of the stomach/Gastric Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy with D2 or greater lymph node dissection
Drug: Gastrectomy+ chemotherapy

SUMMARY:
To evaluate the survival benefit of adjuvant chemotherapy after curative resection with D2 or greater lymph node dissection in T3-4 gastric cancer patients.

DETAILED DESCRIPTION:
Purpose: To evaluate the survival benefit of adjuvant chemotherapy after curative resection in serosa-positive gastric cancer patients, a multicenter phase III clinical trial was conducted by 13 participating centers in Japan. Methods: From January 1993 to March 1998, 268 patients were randomized to either adjuvant chemotherapy (135 pts) or surgery alone (133 pts). The chemotherapy comprised intraperitoneal cisplatin 70 mg/m2 before closing the abdomen, and after surgery intravenous cisplatin 70 mg/m2 (day 14) and 5-fluorouracil (5-FU) 700 mg/m2 daily (day 14-16), and oral FU (UFT) 267 mg/m2 daily from 4 weeks after surgery for the next 12 months. The primary endpoint was overall survival. Relapse-free survival and the site of recurrence were secondary endpoints.

Comparison: gastrectomy with D2 or greater lymph node dissection versus gastrectomy with adjuvant chemotherapy after curative resection in serosa-positive gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Curative operation with D2 or greater lymph node dissection
2. Histologically proven gastric adenocarcinoma
3. Macroscopically serosa-positive (T3-4)
4. No metastases to level 3 - 4 lymph nodes station (N0-2)
5. 75 years or younger
6. Negative peritoneal lavage cytology
7. Adequate organ function WBC >=4000/mm3,Hb >=11.0g/dl,Plt >=100.000/mm3,AST/ALT, T.Bil, BUN, Creatinine <=2.5 x Normal Upper Limit,Creatinine clearance <=70 ml/min
8. Written informed consent

Exclusion Criteria:

1. Prior chemotherapy or radiotherapy
2. Synchronous or metachronous malignancy in other organs

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280
Dates: Start 1993-01; Study Completion 2004-03

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Relapse-free survival
the site of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Furukawa, MD, PhD, Study Chair — Sakai Municipal Hospital
Locations (1):
- Gastric Surgery Division, National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Miyashiro I, Furukawa H, Sasako M, Yamamoto S, Nashimoto A, Nakajima T, Kinoshita T, Kobayashi O, Arai K; Gastric Cancer Surgical Study Group in the Japan Clinical Oncology Group. Randomized clinical trial of adjuvant chemotherapy with intraperitoneal and intravenous cisplatin followed by oral fluorouracil (UFT) in serosa-positive gastric cancer versus curative resection alone: final results of the Japan Clinical Oncology Group trial JCOG9206-2. Gastric Cancer. 2011 Aug;14(3):212-8. doi: 10.1007/s10120-011-0027-3. Epub 2011 Feb 19. PMID 21336855
- See also: Related Info — http://www.jcog.jp/